CLINICAL TRIAL: NCT05999422
Title: Comparison of Exercise Capacity, Physical Activity Level and Quality of Life of Children With Primary Immunodeficiency With Healthy Children
Brief Title: Exercise Capacity, Physical Activity Level and Quality of Life in Children With Primary Immunodeficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof. Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: Gazi University 55
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Primary Immunodeficiency Diseases
Keywords: Primary Immunodeficiency Diseases; Exercise capacity; Quality of life; Physical activity levels
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with primary immunodeficiency: Maximal exercise capacity measured with Cardiopulmonary exercise testing, functional exercise capacity with six minute walk test, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, muscle oxygenation using Moxy monitor, respiratory muscle endurance using incremental threshold loading test, life quality using "Pediatric Quality of Life Inventory™ 4.0 (PedsQL™ 4.0)" (Turkish version).
- Healthy control: Maximal exercise capacity measured with Cardiopulmonary exercise testing, functional exercise capacity with six minute walk test, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, muscle oxygenation using Moxy monitor, respiratory muscle endurance using incremental threshold loading test, life quality using "Pediatric Quality of Life Inventory™ 4.0 (PedsQL™ 4.0)" (Turkish version).

SUMMARY:
This study aims to compare the maximal exercise capacity, functional exercise capacity, respiratory functions, physical activity level, quality of life, respiratory muscle strength and endurance, peripheral muscle strength, muscle oxygenation and dyspnea in children with primary immunodeficiency (PID) and healthy individuals. The study was designed as a cross-sectional study on 26 patients diagnosed with primary immunodeficiency and 26 age- and sex-matched healthy individuals. Differences between both groups will be evaluated statistically. The results of this study aim to reveal how primary immunodeficiency patients are affected by factors such as respiratory functions, physical activity level and quality of life

DETAILED DESCRIPTION:
Primary immune deficiencies (PIDs) are a heterogeneous group of diseases resulting from various abnormalities that affect the development, differentiation, and/or function of cells and components of the immune system. PIDs are clinically characterized by increased susceptibility to infections, autoimmune diseases, auto-inflammatory disorders, allergies, bone marrow failure, and/or malignancies. Although individually rare, the total number of individuals with PIDs constitutes a significant health burden. The prevalence and distribution of PIDs vary among populations, with an estimated prevalence of 1/1,000 to 1/5,000. The specific prevalence of PIDs in Turkey is not well known due to the lack of extensive studies and a national registry system. However, a study encompassing two centers in Turkey reported a prevalence of 30.5/100,000. Currently, approximately 500 PID diseases have been identified, with selective immunoglobulin A (IgA) deficiency being the most common and common variable immunodeficiency (CVID) being the most common symptomatic PID.

Pulmonary complications are highly prevalent among PID patients and significantly contribute to morbidity and mortality. Recurrent respiratory tract infections often serve as the initial warning sign in some PIDs and are a leading cause of mortality in adult PID patients. The presence of two or more pneumonia episodes per year is considered one of the ten warning signs of PID. Acute and chronic infections primarily constitute respiratory system diseases, while non-infectious respiratory complications include asthma, bronchiectasis, bronchiolitis obliterans, interstitial lung disease, granulomatous lung disease, and malignancies. These diseases significantly impact the quality of life of PID patients, limit their working abilities, and restrict their physical and social activities. Health-related quality of life in PID patients is also significantly affected by delays in the diagnosis and treatment of infections.

As survival from infections improves, non-infectious pulmonary complications become more common in PID patients. Particularly in PIDs characterized by antibody deficiencies, permanent lung damage is observed in 20-40% of patients.

Physical activity levels are also affected in PID patients, but there are only survey studies on this topic. Therefore, it is expected that respiratory muscle strength, as well as respiratory muscle endurance, functional exercise capacity, and peripheral muscle strength, would be affected in these patients. There is no research available on maximal exercise capacity, functional exercise capacity, respiratory muscle strength and endurance, and peripheral muscle strength.

The aim of this study is to compare the maximal exercise capacity, functional exercise capacity, respiratory functions, physical activity level, quality of life, respiratory muscle strength and endurance, peripheral muscle strength, muscle oxygenation and dyspnea in patients with primary immune deficiencies with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Individuals aged 6-18 years, diagnosed with primary immune deficiency disease and receiving standard medical treatment, will be included in the study.

Healthy controls:

* Individuals between the ages of 6 and 18 without a known chronic disease will be included.

Exclusion Criteria:

Patients:

* Patients who are uncooperative, have orthopedic or neurological disorders that will affect their exercise capacity, and have pneumonia or any acute infection during the evaluation will be excluded from the study.

Healthy controls:

* Those with a known chronic disease, uncooperative and orthopedic or neurological disorders that will affect their exercise capacity will not be included.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 26 patients diagnosed with primary immune deficiency will be recruited, together with 26 healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Maximal Exercise capacity | through study completion, an average of 1 year
  Maximal Exercise capacity will be evaluated with Cardiopulmonary Exercise testing. The Cardiopulmonary Exercise Testing will be applied according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Functional exercise capacity | through study completion, an average of 1 year
  Functional exercise capacity will be evaluated with the 6- Minute Walk Test. 6- Minute Walk Test will be applied according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Pulmonary function | through study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be measured according to ATS and ERS criteria. With the device, forced vital capacity (FVC), forced expiratory volume in the first second (FEV1) and FEV1 / FVC will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | through study completion, an average of 1 year
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, peak flow rate (PEF) will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | through study completion, an average of 1 year
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Respiratory muscle endurance | through study completion, an average of 1 year
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test with increased threshold load. The test will start with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80% and 100% every two minutes. Patients will be asked to continue breathing through the device during the whole time. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period will be recorded. If the individual can't breathe 3 consecutive times, the test will be terminated by the physiotherapist. The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Respiratory muscle strength | through study completion, an average of 1 year
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be measured with a portable mouth pressure measuring device according to ATS and ERS criteria.
Peripheral muscle strength | through study completion, an average of 1 year
  Isometric peripheral muscle strength will be measured with a portable hand dynamometer (JTECH Commander, USA). Measurements will be repeated on the shoulder abductors and knee extensors three times on the right and left.
Muscle Oxygenation (Local oxygen saturation (SmO2)) | through study completion, an average of 1 year
  Muscle Oxygenation will be measured with Moxy device monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device will be placed on the motor point of quadriceps muscle during Cardiopulmonary Exercise Testing as well as during the six minute walk test. Local oxygen saturation (SmO2) levels will be measured.
Muscle Oxygenation (Total haemoglobin (THb)) | through study completion, an average of 1 year
  Muscle Oxygenation will be measured with Moxy device monitor (Moxy, Fortiori Design LLC, Minnesota, USA). The device will be placed on the motor point of quadriceps muscle during Cardiopulmonary Exercise Testing as well as during the six minute walk test. Total haemoglobin (THb) levels will be measured.
Physical activity (Total energy expenditure) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity (Physical activity time (min / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Physical activity time (min / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity (Average metabolic equivalent (MET / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity (Number of steps (steps / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity (Time spent lying down (min / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Time spent lying down (min / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical Activity (Sleep time (min / day)) | through study completion, an average of 1 year
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multi sensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient was informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The measured parameter will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Pediatric Quality of Life Inventory™ 4.0 (Quality of Life Questionnaire) | through study completion, an average of 1 year
  The quality of life will be measured with the Turkish version of Pediatric Quality of Life Inventory™ 4.0 (PedsQL™ 4.0). PedsQL measures health related quality of life in children and adolescents. The measure can be completed by parents (the Proxy Report) as well as children and young people (the Self-Report). The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization, as well as role (school) functioning. The four scales that it measures are Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items) and School Functioning (5 items). Each item of the instrument is scored on a 5-point scale. Scale scores are computed as the sum of the items over the number of items answered.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, Prof.Dr., Study Director — Gazi University; Riad Bejta, B.sc PT, Study Chair — Gazi University; Caner Aytekin, Assoc. Prof, Principal Investigator — MH. Dr. Sami Ulus Children's Health and Diseases Training and Research Hospital
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tangye SG, Al-Herz W, Bousfiha A, Cunningham-Rundles C, Franco JL, Holland SM, Klein C, Morio T, Oksenhendler E, Picard C, Puel A, Puck J, Seppanen MRJ, Somech R, Su HC, Sullivan KE, Torgerson TR, Meyts I. Human Inborn Errors of Immunity: 2022 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2022 Oct;42(7):1473-1507. doi: 10.1007/s10875-022-01289-3. Epub 2022 Jun 24. PMID 35748970
- [Background] Tangye SG, Al-Herz W, Bousfiha A, Chatila T, Cunningham-Rundles C, Etzioni A, Franco JL, Holland SM, Klein C, Morio T, Ochs HD, Oksenhendler E, Picard C, Puck J, Torgerson TR, Casanova JL, Sullivan KE. Human Inborn Errors of Immunity: 2019 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2020 Jan;40(1):24-64. doi: 10.1007/s10875-019-00737-x. Epub 2020 Jan 17. PMID 31953710
- [Background] Kilic SS, Ozel M, Hafizoglu D, Karaca NE, Aksu G, Kutukculer N. The prevalences [correction] and patient characteristics of primary immunodeficiency diseases in Turkey--two centers study. J Clin Immunol. 2013 Jan;33(1):74-83. doi: 10.1007/s10875-012-9763-3. Epub 2012 Sep 15. PMID 22983506
- [Background] Ameratunga R, Longhurst H, Lehnert K, Steele R, Edwards ESJ, Woon ST. Are All Primary Immunodeficiency Disorders Inborn Errors of Immunity? Front Immunol. 2021 Jul 21;12:706796. doi: 10.3389/fimmu.2021.706796. eCollection 2021. No abstract available. PMID 34367167
- [Background] Hampson FA, Chandra A, Screaton NJ, Condliffe A, Kumararatne DS, Exley AR, Babar JL. Respiratory disease in common variable immunodeficiency and other primary immunodeficiency disorders. Clin Radiol. 2012 Jun;67(6):587-95. doi: 10.1016/j.crad.2011.10.028. Epub 2012 Jan 9. PMID 22226567
- [Background] Verma N, Grimbacher B, Hurst JR. Lung disease in primary antibody deficiency. Lancet Respir Med. 2015 Aug;3(8):651-60. doi: 10.1016/S2213-2600(15)00202-7. Epub 2015 Jul 15. PMID 26188881
- [Background] Modell V, Orange JS, Quinn J, Modell F. Global report on primary immunodeficiencies: 2018 update from the Jeffrey Modell Centers Network on disease classification, regional trends, treatment modalities, and physician reported outcomes. Immunol Res. 2018 Jun;66(3):367-380. doi: 10.1007/s12026-018-8996-5. PMID 29744770
- [Background] Quinti I, Di Pietro C, Martini H, Pesce AM, Lombardi F, Baumghartner M, Colantuono S, Milito C, Tabolli S. Health related quality of life in common variable immunodeficiency. Yonsei Med J. 2012 May;53(3):603-10. doi: 10.3349/ymj.2012.53.3.603. PMID 22477006
- [Background] Routes J, Costa-Carvalho BT, Grimbacher B, Paris K, Ochs HD, Filipovich A, Hintermeyer M, de Melo KM, Workman S, Ito D, Ye X, Bonnet P, Li-McLeod J. Health-Related Quality of Life and Health Resource Utilization in Patients with Primary Immunodeficiency Disease Prior to and Following 12 Months of Immunoglobulin G Treatment. J Clin Immunol. 2016 Jul;36(5):450-61. doi: 10.1007/s10875-016-0279-0. Epub 2016 Apr 18. PMID 27091140
- [Background] Urschel S, Kayikci L, Wintergerst U, Notheis G, Jansson A, Belohradsky BH. Common variable immunodeficiency disorders in children: delayed diagnosis despite typical clinical presentation. J Pediatr. 2009 Jun;154(6):888-94. doi: 10.1016/j.jpeds.2008.12.020. Epub 2009 Feb 23. PMID 19230900
- [Background] Jesenak M, Banovcin P, Jesenakova B, Babusikova E. Pulmonary manifestations of primary immunodeficiency disorders in children. Front Pediatr. 2014 Jul 25;2:77. doi: 10.3389/fped.2014.00077. eCollection 2014. PMID 25121077
- [Background] Azizi G, Abolhassani H, Asgardoon MH, Alinia T, Yazdani R, Mohammadi J, Rezaei N, Ochs HD, Aghamohammadi A. Autoimmunity in common variable immunodeficiency: epidemiology, pathophysiology and management. Expert Rev Clin Immunol. 2017 Feb;13(2):101-115. doi: 10.1080/1744666X.2016.1224664. Epub 2016 Sep 16. PMID 27636680
- [Background] Manson D, Reid B, Dalal I, Roifman CM. Clinical utility of high-resolution pulmonary computed tomography in children with antibody deficiency disorders. Pediatr Radiol. 1997 Oct;27(10):794-8. doi: 10.1007/s002470050235. PMID 9323243
- [Background] Sowers KL, Litwin BA, Lee ACW, Galantino MLA. Exercise Perception and Behaviors in Individuals Living with Primary Immunodeficiency Disease. J Clin Immunol. 2018 Feb;38(2):174-184. doi: 10.1007/s10875-017-0472-9. Epub 2018 Jan 6. PMID 29307028